CLINICAL TRIAL: NCT02443935
Title: Toll-like Receptor 9 Enhancement of Antiviral Immunity in Chronic HIV-1 Infection: a Phase 1b/2a Trial
Brief Title: Toll-like Receptor 9 Agonist Treatment in Chronic HIV-1 Infection
Acronym: TEACH
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TEA-001
Record Dates: First submitted 2015-04-30; First posted 2015-05-14 (Estimated); Last update posted 2017-06-29 (Actual); Status verified 2015-04

CONDITIONS: HIV
MeSH Terms: interventions — MGN1703

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MGN1703 (Experimental): TLR-9 agonist MGN1703 administered to HIV-1 positive patients on cART
  Interventions: Drug: MGN1703

INTERVENTIONS:
Drug: MGN1703 — 60 mg s.c. twice weekly for 4 weeks
  Other Names: TLR9 agonist; CpG oligodeoxynucleotides
Drug: MGN1703 — 60 mg s.c. twice weekly for 24 weeks
  Other Names: TLR9 agonist; CpG oligodeoxynucleotides

SUMMARY:
Combination antiretroviral treatment (cART) effectively suppresses virus replication and partially restores immune functions. However, cART cannot cure HIV infection.

This study aim to investigate whether the antiviral immune response can be enhanced and/or viral transcription reactivated with MGN1703. MGN1703 is an agonist to toll-like receptor (TLR) 9. Activation of TLR9 has been shown to augment innate and adaptive immune effector functions, most notably enhanced NK cell and T cell functions.

Furthermore, TLR9 agonists have been shown in vitro to reactivate viral transcription in latently infected cells, potentially leading to enhanced recognition of infected cells by the immune effector cells.

DETAILED DESCRIPTION:
In Part A, participants will receive 4 weeks MGN1703 therapy (60 mg s.c. twice weekly). During the 4 weeks, participants will be closely monitored for safety and therapeutic effects of the drug. Targeted enrolment in Part A is 14-16 study subjects.

In Part B, participants will receive 24 weeks of MGN1703 therapy (60 mg s.c. twice weekly). During the 24 weeks, participants will be frequently monitored for safety and therapeutic effects of the drug. Targeted enrolment in Part B is 10-12 study subjects, preferentially recruited from part A.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 infection
* Age >18 years
* CD4+ T-cell count >350/µL at screening
* On cART (for a minimum of 12 months)
* Able to give informed consent.

Exclusion Criteria:

* Pregnancy as determined by a positive urine beta-hCG (if female)
* Males or females who are unwilling or unable to use barrier contraception during sexual intercourse for the entire study period.
* Currently breast-feeding (if female)
* Viral load (HIV RNA) > 50 copies/mL
* Contraindication to receive MGN1703 as per current investigator brochure
* Presence of acute bacterial infection or undiagnosed febrile condition
* Concurrent chronic systemic immune therapy or immunosuppressant medication, including continuous systemic steroid treatment within the last 2 weeks prior to randomization
* Use of antibiotic therapy within the last 2 weeks prior to randomization
* Known HBV or HCV infection
* Any medical, psychiatric, social, or occupational condition or other responsibility that, in the judgment of the Principal Investigator (PI), would interfere with the evaluation of study objectives (such as severe alcohol abuse, severe drug abuse, dementia)
* Unable to follow protocol regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-04; Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-25 (Actual)

PRIMARY OUTCOMES:
Part A: NK cell activation | 12 weeks
  As measured by CD69 expression
Part B: Quantification of the size of the HIV reservoir | 32 weeks
  As measured by quantitative viral outgrowth (qVOA) and total HIV DNA

SECONDARY OUTCOMES:
Safety and tolerability, as measured by adverse events (AE), adverse reactions (AR), serious adverse events (SAE), serious adverse reactions (SAR) and suspected unexpected serious adverse reactions (SUSAR). | 12 weeks
  Safety evaluation, as measured by adverse events (AE), adverse reactions (AR), serious adverse events (SAE), serious adverse reactions (SAR) and suspected unexpected serious adverse reactions (SUSAR).
The size of the HIV-1 reservoir | 12 weeks
  HIV DNA and others measures
Viral transcription | 12 weeks
  Plasma HIV RNA and cell-associated unspliced HIV RNA

OTHER OUTCOMES:
Effects of MGN1703 on T and NK cell activation in the gut | 12 weeks
  Changes in the expression of activation markers such as CD69.

CONTACTS AND LOCATIONS:
Overall Officials: Lars J Østergaard, MD,PhD,DMSc, Study Chair — Department for Infectious Diseases, Aarhus University Hospital, Denmark
Locations (2):
- Denmark (2):
  - Department for Infectious Diseases, Aarhus University Hospital, Aarhus N
  - Department for Infectious Diseases, Amager and Hvidovre Hospitals, Hvidovre

REFERENCES:
- [Derived] Vibholm LK, Konrad CV, Schleimann MH, Frattari G, Winckelmann A, Klastrup V, Jensen NM, Jensen SS, Schmidt M, Wittig B, Zuwala K, Mack K, Olesen R, Hua S, Lichterfeld M, Ostergaard L, Denton PW, Tolstrup M, Sogaard OS. Effects of 24-week Toll-like receptor 9 agonist treatment in HIV type 1+ individuals. AIDS. 2019 Jul 1;33(8):1315-1325. doi: 10.1097/QAD.0000000000002213. PMID 30932955
- [Derived] Vibholm L, Schleimann MH, Hojen JF, Benfield T, Offersen R, Rasmussen K, Olesen R, Dige A, Agnholt J, Grau J, Buzon M, Wittig B, Lichterfeld M, Petersen AM, Deng X, Abdel-Mohsen M, Pillai SK, Rutsaert S, Trypsteen W, De Spiegelaere W, Vandekerchove L, Ostergaard L, Rasmussen TA, Denton PW, Tolstrup M, Sogaard OS. Short-Course Toll-Like Receptor 9 Agonist Treatment Impacts Innate Immunity and Plasma Viremia in Individuals With Human Immunodeficiency Virus Infection. Clin Infect Dis. 2017 Jun 15;64(12):1686-1695. doi: 10.1093/cid/cix201. PMID 28329286